CLINICAL TRIAL: NCT07190560
Title: Against Chikungunya Virus and Neonatal Infection
Acronym: ConvictionCHIK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/RUN/0036
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chikungunya Virus Infection; Neonatal; Transfusion; Encephalopathy
MeSH Terms: conditions — Chikungunya Fever; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma transfusion in newborns whose mothers are infected with chikungunya around the time of birth. (Experimental): Biological and medical examination from Day 1 to Day 7 and at a visit between 1 and 3 months
  Interventions: Biological: plasma transfusion : PC-CHIK-V
- Parallel observational cohort (No Intervention): No intervention, secondary using of care data collected, during standard cares, for the research

INTERVENTIONS:
Biological: plasma transfusion : PC-CHIK-V — plasma transfusion , from donation from an individual who has declared a Chikungunya infection for less than 6 months , to a newborn, whose mother has a peripartum chikungunya infection
  Arms: Plasma transfusion in newborns whose mothers are infected with chikungunya around the time of birth.

SUMMARY:
The goal of this clinical trial is to learn if administration of plasma, from a whole blood donation from an individual who has declared a Chikungunya infection for less than 6 months , to a newborn, whose mother has a peripartum chikungunya infection, will have an impact on the proportion of newborns surviving without encephalitis/encephalopathy (EE) within the first 5 days of life. Researchers will compare results to an observational study of 30 newborns who couldn't have been proposed to participate at the clinical trial, because of delay of diagnosis or delay of transfer to hospital which doesn't allow transfusion or parents not accepting plasma transfusion to the newborn.

Participants of the clinical trial will:

* receive a transfusion,
* visit the clinic and undergo biological tests every day until day 7 and once between 1 and 3 months.

Participant of observational study as part of their regular medical care, and biological data will be reused for the research from the mother's diagnosis until the newborn reaches 3 months of age

ELIGIBILITY:
Inclusion Criteria:

* Treatment group

Newborn:

* whose mother has a clinical and/or laboratory diagnosis of Chikungunya (CHIK) infection occurring between 2 days before and 2 days after birth.
* Hospitalized in a Level III neonatology unit in Mayotte or at the University Hospital of La Réunion.
* Eligible for experimental treatment (called PC-CHIK-V):

  * If the maternal infection was diagnosed between2 days before and the day of delivery, treatment can be administered within the first 12 hours of the newborn's life.
  * If the maternal infection was diagnosed between 1 day and 2 days after birth, treatment can be administered within 12 hours of diagnosis.
* Whose holders of parental authority have given free, informed, and written consent prior to any examination required for the research. Parallel Cohort of

Untreated Newborns (parallel observational cohort)

Newborns:

* Whose mother has a clinical and/or laboratory diagnosis of CHIK-V infection occurring between 2 days before and 2 days after birth.
* Hospitalized in a Level III neonatology unit in Mayotte or at the University Hospital of La Réunion.
* Not treated with PC-CHIK-V:
* Monitored in one of the units of the Neonatology Department for at least 5 days from the day of birth.
* Whose holders of parental authority (or the holder if the mother is the sole holder of parental authority) have been informed of the research and have not objected to the use of data collected during hospitalization for research purposes.

Exclusion Criteria:

* Newborns who present at birth with clinical criteria for ahypoxic-ischemic encephalopathy (HIE) that require therapeutic hypothermia according to the national protocol for "neonatal therapeutic hypothermia"
* Newborns who require phototherapy treatment at the time of enrollment using devices with a maximum energy wavelength less than 425 nm and/or with an emission bandwidth with a lower limit of <375 nm.

Ages: 0 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of early administration of PC-CHIK-V in preventing the occurrence of neonatal CHIK-V encephalitis/encephalopathy (EE) in newborns whose mothers have peripartum CHIK-V infection. | Five days after inclusion
  The primary outcome measure is the proportion of newborns treated with PC-CHIK-V surviving without encephalitis/encephalopathy (EE) within the first 5 days of life.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU La Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: Undecided